CLINICAL TRIAL: NCT04740554
Title: Characterization of Heart Rate Variability in Individuals With Duchenne Muscular Dystrophy - Influence of Corticosteroids and Betablockers
Brief Title: Heart Rate Variability in Individuals With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Researcher, University of Sao Paulo
Other Study IDs: 09942913.4.0000.5505
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Muscular Dystrophy, Duchenne; Prednisone; Deflazacort
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — deflazacort; Prednisone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Duchenne Muscular Dystrophy group with Deflazacort: Individuals Duchenne Muscular Dystrophy, with age 11 to 18 years which make use of deflazacort.
  Interventions: Behavioral: Duchenne Muscular Dystrophy group with Deflazacort
- Duchenne Muscular Dystrophy group with Prednisone/Predisolone: Individuals Duchenne Muscular Dystrophy, with age 11 to 18 years which make use of Prednisone/Predinisolone.
  Interventions: Behavioral: Duchenne Muscular Dystrophy group with Prednisone/Predisolone
- Duchenne Muscular Dystrophy group without Corticosteroids therapy: Individuals Duchenne Muscular Dystrophy, with age 11 to 18 years which don't use of corticosteroids.
  Interventions: Behavioral: Duchenne Muscular Dystrophy group without Corticosteroids therapy
- Control Group Typically Developing: Individuals with typical development age 11 to 18 years which don't use of corticosteroids.
  Interventions: Behavioral: Control Group Typically Developing

INTERVENTIONS:
Behavioral: Duchenne Muscular Dystrophy group with Deflazacort — Subjects with duchenne muscular dystrophy undergoing drug therapy with Deflazacort
  Groups: Duchenne Muscular Dystrophy group with Deflazacort
Behavioral: Duchenne Muscular Dystrophy group with Prednisone/Predisolone — Subjects with duchenne muscular dystrophy undergoing drug therapy with Prednisona/Predinisolone
  Groups: Duchenne Muscular Dystrophy group with Prednisone/Predisolone
Behavioral: Duchenne Muscular Dystrophy group without Corticosteroids therapy — Control group with duchenne muscular dystrophy without the use of corticosteroid drug therapy.
  Groups: Duchenne Muscular Dystrophy group without Corticosteroids therapy
Behavioral: Control Group Typically Developing — Control group with tipical development.
  Groups: Control Group Typically Developing

SUMMARY:
A cross-sectional study was carried out, in which 40 boys, aged 11 to 18 years, were evaluated. The recruitment of groups was carried out at the neuromuscular disease outpatient clinic of the Federal University of São Paulo (UNIFESP). The recruited individuals were divided into 4 groups, namely: DMD that used deflazacort (DMD-D); DMD that used Prednisone/Prednisolone (DMD-P); DMD Control with no corticoid use (DMD-C) and Controls with typical development (CTD). The protocol was applied during the evaluation that was carried out at outpatient follow-up visits.

To assess the functionality of each patient, the Vignos scales were used to characterize the sample and the Motor Function Measure (MFM) for association with HRV indices.

All heart rate records were performed using a cardiofrequencymeter (V800, Polar). After placing the brace and monitor, the individuals were placed in the supine position and remained at rest spontaneously breathing for 25 minutes. For HRV analysis, indexes obtained by linear methods, in the domain of time and frequency, and non-linear methods were used.

DETAILED DESCRIPTION:
A cross-sectional study was carried out, in which 40 boys, aged 11 to 18 years, were evaluated. The recruitment of groups was carried out at the neuromuscular disease outpatient clinic of the Federal University of São Paulo (UNIFESP). The recruited individuals were divided into 4 groups, namely: DMD that used deflazacort (DMD-D) with n=11; DMD that used Prednisone/Prednisolone (DMD-P), with n=9; DMD Control with no corticoid use (DMD-C), and n=10 and Controls with typical development (CTD) with n=10. The protocol was applied during the evaluation that was carried out at outpatient follow-up visits. Anthropometry was analyzed in 4 groups and functionality was assessed in 3 groups with DMD. To assess the functionality of each patient, the Vignos scales were used to characterize the sample and the Motor Function Measure (MFM) for association with HRV indices.

Initially, the resting ECG was analyzed to verify the existence of sinus rhythm and to exclude individuals with arrhythmias and blocks. The measurements at rest were performed immediately before and after the HRV assessment, including systolic (SBP) and diastolic (DBP), heart rate (HR), Respiratory Rate (RF - blood pressure) to ensure that at the beginning and at the end of the collection FR remains between 9 - 24rpm, in the range of 0.15 - 0.40Hz) and partial oxygen saturation (SO2). Heart rate was recorded by the cardiofrequency meter (RS800CX, Polar). And the partial oxygen saturation by means of a digital oximeter (DX2010, Dixtal) connected to the participant's index finger or hallux, through a sensor of age-appropriate size, in room air. Hemoglobin saturation by oxygen was recorded after the first minute of stabilization, as the value that remains most constant during the second minute.

All heart rate records were performed using a cardiofrequencymeter (V800, Polar). After placing the brace and monitor, the individuals were placed in the supine position and remained at rest spontaneously breathing for 25 minutes. For HRV analysis, indexes obtained by linear methods, in the domain of time and frequency, and non-linear methods were used.

In the time domain, for linear analyses, each normal RR interval (sinus beats) was verified during a certain time interval and, using statistical and non-linear methods, the translating indexes of fluctuations in the duration of the cardiac cycles were calculated. With this, the indices expressed in ms were obtained: SDNN (Standard deviation of the normal RR intervals recorded in a time interval); rMSSD (square root of the mean of the square of the differences between adjacent normal RR intervals in a time interval).

In the frequency domain, the spectral power density is more used, mainly when treating individuals in resting conditions. This analysis divides HRV into fundamental oscillatory components, which were used the main: High Frequency normalized unite (HFnu) component and Low Frequency normalized unite (LFnu) component. O algoritmo utilizado para a análise espectral foi a transformada rápida de Fourier - FFT (janela de 256 s com 50% de overlap).

Among the nonlinear methods used for HRV analysis, we can mention the Detrended Fluctuations Analysis (DFA), Visual Recurrence Analysis (VRA) and symbolic analysis (SA), the three of which were verified in this study.

DFA is used to quantify the fractal property of RR interval time series, being used to detect possible abnormalities present in a subject, based on α coefficients. For this, short memory parameters α1, which corresponds to a period of 4 to 11 beats, and long memory α2, which corresponds to the period from 64 to 1024 beats, were used.

The VRA is used to study the time dependence of a series, that is, in the study of stationarity35. The recurrence graph makes it possible to visualize the behavior of trajectories in the phase space and, in addition, to show the times in which a state of a dynamic system is repeated, besides these factors can be confirmed regarding the quantitative analysis of this, wich presents such indices: Mean, SD, PerRec, PerDet, PerLam, TrapTim, Ratio.

The evaluation of the symbolic analysis is based on the quantification of the information carried in a time series, in the transformation of the previously selected iRRs into integers from zero to six, from which sequences of 3 symbols (symbolic patterns) are constructed. For this, all possible patterns will be grouped according to the number and type of variations between the symbols, shown subsequently. The patterns were (1) patterns, without variation (0V), three identical symbols; (2) patterns with a variation (1V), that is, two subsequent symbols that are the same and a different one; (3) patterns with two similar variations (2LV) that is, the three symbols form a ramp; (4) patterns with two different variations (2ULV), that is, the three symbols form a peak or a valley.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with DMD confirmed by molecular method and / or by protein expression of skeletal muscle.
* Individuals undergoing clinical follow-up at the outpatient clinic for neuromuscular diseases at the Federal University of São Paulo (UNIFESP)
* Individuals who had authorization from their parents or guardians to participate in the study

Exclusion Criteria:

* Patients with cardiac arrhythmias.
* Patients with atrioventricular block.
* Patients with congenital anomalies such as congenital heart defects, pulmonary deformity.
* Patients using drugs that interfere with ANS, such as antiarrhythmic agents and drugs for the treatment of diabetes mellitus, such as insulin.

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — It is a disease that affects only male
Study Population: 30 boys with Duchenne Muscular Dystrophy and 10 typically developing boys aged 11 to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability in adolescents with Duchenne Muscular Dystrophy undergoing therapy with corticosteroids | One day
  Heart rate variability indices at rest in adolescents with duchenne muscular dystrophy will be analyzed, which will be divided into the following groups: Under the use of Deflazacort, Predinisone / Predinisolone and without the use of corticosteroids, in addition to the analysis of a control group with typical development.

CONTACTS AND LOCATIONS:
Overall Officials: Talita D da Silva, Ph.D., Principal Investigator — Universidade Federal de São Paulo

IPD SHARING:
Plan to Share IPD: No